CLINICAL TRIAL: NCT06523582
Title: Genetic Bases of Neuroendocrine Neoplasms in Mexican Patients
Status: Recruiting | Type: Observational
Sponsor: Universidad Nacional Autonoma de Mexico (Other)
Collaborators: Instituto Mexicano del Seguro Social (Other Government); Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Laura Cristina Hernández Ramírez, Associate Researcher C, Universidad Nacional Autonoma de Mexico
Other Study IDs: IMSSR-2022-785-011/INCMNSZ4090
Record Dates: First submitted 2024-07-17; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Neuroendocrine Neoplasm; Neuroendocrine Neoplasm of Gastrointestinal Tract; Neuroendocrine Neoplasm of Lung; Thymic Neuroendocrine Neoplasm; Neuroendocrine Tumor of Pancreas; Gastrointestinal Stromal Tumors; Medullary Thyroid Cancer; Paraganglioma; Pheochromocytoma; Primary Hyperparathyroidism; Pituitary Tumor; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia Type 2; Multiple Endocrine Neoplasia Type 4; Carney Complex; Carney Stratakis Dyad; Carney Triad; Cowden Syndrome; DICER1 Syndrome; Li-Fraumeni Syndrome; Lynch Syndrome; Von Hippel-Lindau Disease; Familial Isolated Pituitary Adenoma; X-Linked Acrogigantism; Neurofibromatosis 1; Tuberous Sclerosis
MeSH Terms: conditions — Neuroendocrine Tumors; Adenoma, Islet Cell; Gastrointestinal Stromal Tumors; Carcinoma, Medullary; Paraganglioma; Pheochromocytoma; Hyperparathyroidism, Primary; Pituitary Neoplasms; Multiple Endocrine Neoplasia Type 1; Multiple Endocrine Neoplasia Type 2a; Carney Complex; Carney-Stratakis Syndrome; Carney Triad; Hamartoma Syndrome, Multiple; Li-Fraumeni Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; von Hippel-Lindau Disease; Pituitary Adenoma, Familial Isolated; Neurofibromatosis 1; Tuberous Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A 5 ml sample of peripheral blood obtained by phlebotomy will be collected in a tube with EDTA at recruitment and stored at 4°C until processing. Archival formalin-fixed paraffin-embedded tissues samples will be obtained for patients with previous tumor resection, and fresh frozen tissue samples will be obtained por individuals undergoing surgical tumor excision in the course of the study, when possible. DNA, and in selected cases, RNA, will be extracted from blood and tissue samples and will be stored at -20 °C or -80 °C, respectively, for the durantion of the study. A unique deidentified code for each participant will be used for sample labelling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neuroendocrine neoplasms (NENs) are a heterogeneous group of lesions derived from cells with the ability to produce hormones that may arise from multiple different organs. Their clinical behavior is quite variable, encompassing both benign lesions and aggressive tumors that invade surrounding and/or distant structures. NENs may also cause serious morbidity due to hormone oversecretion. NENs are among the most frequently inherited human tumors, presenting either isolated or as part of syndromes in which a single patient or family develops multiple tumors. There are also non-inherited changes in the genetic information of the tumor cells that are potential targets for treatment. Both inherited and non-inherited DNA defects can be identified using modern routine genetic tests which, unfortunately, are not widely available in Mexico.

This project seeks to uncover the genetic defects causing NENs in a large cohort of Mexican patients, using three different methods for genetic testing. Adult individuals with various types of NENs from two reference hospitals in Mexico City will be invited to participate. After completing informed consent, blood and, if possible, tissue samples will be obtained from all participants. Clinical details, laboratory results, imaging studies, and histopathological data at disease presentation will be retrieved.

An initial screening will be performed by analyzing changes in the sequence of multiple genes that have been associated with the occurrence of NENs. In cases with negative screening, a specific method to assess changes in the number of copies of the same genes will also be employed. Finally, sequences of all DNA regions encoding information required to make proteins will be obtained in selected cases. Analyses will be carried out in blood and, if available, also in tumor tissue samples from study participants. Screening of additional family members will be offered.

This project will accurately describe the repertoire of specific defects causing NENs in the study population, and will likely uncover and characterize novel genetic associations. The results will contribute for a better understanding of the alterations within and outside known driver genes that shape syndromic presentations, tumor behaviors, and inheritance patterns in individuals with NENs. These data will contribute to improve the information on the molecular bases of NENs, including alterations that can be used as therapeutic targets.

DETAILED DESCRIPTION:
Introduction.

NENs are a heterogeneous group of human neoplasms with a variable clinical behavior, spanning from indolence to frank aggressiveness and malignancy. They arise from various tissues with common embryological origins that share the capacity for producing hormones. Their growth might compromise surrounding structures and they often cause significant morbidity due to their associated syndromes of hormone oversecretion. Although traditionally considered rare, the frequency of NENs has greatly increased in the last decades, due to improved clinical awareness and diagnostic strategies. This group includes lesions such as bronchopulmonary, gastrointestinal, pancreatic, and thymic NENs, medullary thyroid carcinoma (MTC), paragangliomas and pheochromocytomas (PPGLs), parathyroid adenomas and carcinomas, and pituitary neuroendocrine tumors (PitNETs), among others.

Interestingly, NENs are among the human neoplasms with a strongest heritable component. Some NENs are part of autosomal dominant syndromes of multiple endocrine neoplasia, where they present in combination with other characteristic endocrine and non-endocrine tumors in the same individual and/or family. Clinical descriptions of such entities exist in the literature since the mid-twentieth Century, although their genetic causes were not determined until three or four decades ago. In other instances, a single type of tumor, such as MTC, PitNETs, or PPGLs, arises in multiple members of the same family, without other associated features. Occasionally, individuals with apparently sporadic presentation are indeed simplex cases of familial conditions. It is currently known that around 50% of cases of MTC, 40% of PPGLs, 20% of gastrointestinal, pancreatic, bronchopulmonary, and thymic NENs, 15% of parathyroid NENs, and 5-10% of PitNETs are due to germline defects. Aside from heritable genetic defects, alterations at the somatic level determine specific clinical courses in both sporadic and familial NENs.

In the last decade, the widespread use of powerful tools for genetic analyses has resulted in a dramatic increase in the known genetic causes of NENs. These approaches have also yielded previously unsuspected genotype-phenotype associations and have uncovered a great overlap in the clinical presentation of different syndromes of multiple endocrine neoplasia. Genetic tests are key for early diagnosis, tailored clinical management, and genetic counseling. Moreover, genetic analyses on the tumors have uncovered potential biomarkers and therapeutic targets. Yet, platforms for genetic diagnosis are not widely available and data on genetic disease drivers do not accurately represent all human populations. Genetic tests are not widely available in Mexico and are almost non-existent in its public hospitals, which serve the majority of the country's ∼128 million population. Interestingly, Mestizos, which account for most of the Mexican population, are one of the most genetically diverse human groups. Precision medicine strategies require population-specific information, yet, Mexican Mestizos are poorly represented in international genetic databases.

Aims.

Using a precise, robust, and affordable testing platform, this project will describe the repertoire and frequency of germline and somatic genetic causes of NENs in a large prospective cohort of Mexican Mestizos. It will also define the phenotypes and clinical outcomes associated with specific genetic defects and explore the functional consequences of new defects in genes previously associated with these neoplasms. Finally, it will uncover and thoroughly characterize novel genetic associations, including potential druggable targets.

Methods.

Approval for the study has been obtained from the Institutional Review Boards of two reference hospitals: Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán (INCMNSZ, project 4090), and Hospital de Especialidades de Centro Médico Nacional Siglo XXI, Instituto Mexicano del Seguro Social (IMSS, project R-2022-785-011). Under informed consent, DNA samples from blood and fresh or formalin-fixed and paraffin-embedded tumors will be obtained. All experimental methods, except exome sequencing, will be carried out at the Research Support Network of the Universidad Nacional Autónoma de México and INCMNSZ. The study started in August 2022 and is designed as a 15-year prospective cohort with an estimated total of 750 participants. Adult individuals (age ≥18 years at recruitment) with new or previous diagnosis of any type of NEN will be invited to participate, including sporadic, familial, isolated, and syndromic presentations. All participants will be offered the opportunity to obtain the results of their genetic studies. A unique deidentified code will be used to label all samples and data collected for each participant, to protect their personal information.

Details on family history, clinical presentation, biochemical, imaging, histopathological, and previous genetic studies for each participant will be entered into a deidentified electronic clinical database. Data on clinical outcomes will be collected prospectively for a maximum of 15 years. For all cases, a 5 ml peripheral blood sample will be collected in a tube with EDTA at recruitment and stored at 4°C until processing. DNA will be extracted from blood samples within 24 h after collection. Archival formalin-fixed paraffin-embedded (FFPE) tissue samples will be obtained for patients with previous tumor resection, when available. When possible and without interfering with routine histopathological analyses, fresh frozen tissue samples will be obtained from individuals undergoing surgical tumor excision in the course of the study. Frozen tissues will be stored in liquid nitrogen until processing. DNA will be extracted from all tissue samples and RNA will be extracted from blood or tissue samples in selected cases. Sample quality and concentration will be analyzed by spectrophotometry and fluorometry. DNA will be stored at -20 °C and RNA will be stored at -80 °C for the duration of the study.

DNA samples will be analyzed using multiple techniques, consisting of a first step of targeted next generation sequencing (NGS), followed by targeted array-based comparative genomic hybridization (aCGH) and exome sequencing (ES). For NGS, a customized panel including 54 genes with a known association with NENs has been designed, using the Twist Biosciences platform. Libraries from blood DNA from all participants and, when possible, fresh tumor DNA, will be prepared according to the manufacturer's instructions and sequenced in an Illumina MiSeq instrument at an approximate depth of 300x. Sequences will be mapped to the GRCh38/hg38 human genome, PCR duplicates will be marked, and variant calling will be carried out for single nucleotide variants (SNVs), indels, and copy number variants. Variants will be selected based on their frequency (<0.1% in both general population and Mexican population databases), previous classification (according to the American College of Medical Genetics and Genomics and Association for Molecular Pathology guidelines) reported in ClinVar, results from multiple in silico prediction tools, and literature search for additional clinical and experimental data.

For selected cases remaining without genetic diagnosis after the NGS panel, CNV analysis of the same targeted regions will be carried out. For this purpose, a high density aCGH targeting the same regions of interest than the NGS panel has been designed, using the Agilent SureDesign platform. Samples will be processed in a 16 x 25 K array format and the results will be analyzed with the Agilent Genomic Workbench software. Variant filtering and classification will be done in a similar manner as described for SNVs and indels.

All relevant variants classified as pathogenic and likely pathogenic will be subjected to orthogonal validation (Sanger sequencing for SNVs and indels and droplet digital polymerase chain reaction for CNVs). All participants choosing to know their results will receive detailed reports including all relevant variants of uncertain significance (VUS), as well as likely pathogenic, and pathogenic variants with an interpretation of their clinical significance. When clinically indicated, participants will be offered cascade targeted screening of additional family members. Selected VUS, including variants not previously reported, will be subjected to additional evaluations, including search for loss of heterozygosity in tumor tissues, expression assays, coding DNA sequencing and/or breakpoint analyses in blood and/or tumor tissues, or experimental functional validation.

The genetic results will be correlated with the clinical data to determine the frequency and type of genetic defects associated to each phenotype in the study population. Conversely, thorough clinical descriptions of the repertoire of phenotypes associated with each specific genetic defect will be obtained. The influence of particular genotype-phenotype associations on the clinical presentation and clinical outcomes will also be explored. Cases with no genetic diagnosis after targeted NGS and aCGH will be subjected to exome sequencing. Groups of patients with similar phenotypes will be analyzed together to identify disease-specific defects in genes not previously associated with NENs. Novel candidate associations will be thoroughly characterized using custom-designed combinations of experimental approaches plus additional screening in affected families.

Expected results.

Incorporating multiple phenotypes of NENs in the proposed novel platform for general genotyping will significantly improve the probability of variant detection, compared with the currently available genetic tests. In addition to generating a large amount of genetic and clinical data for previously unexplored phenotypes in the study population, this project will very likely also identify novel disease modifiers and founder variants. These data will contribute to the development of population- and genotype-specific strategies for genetic counseling, early diagnosis, clinical follow up, and treatment, thereby improving the future outcomes of individuals with NENs. This strategy will uncover the landscape of germline and somatic NEN-associated defects in an extremely genetically diverse population that is poorly represented in international studies. The results will be compared with data from other populations to better understand the alterations within and outside known driver genes that shape syndromic presentations, tumor behaviors, and inheritance patterns in NENs.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with a new or previous clinical diagnosis of any of the following conditions:

* Isolated NENs with sporadic presentation, including bronchopulmonary NENs, gastrointestinal NENs, medullary thyroid carcinoma, pancreatic NENs, paragangliomas, pheochromocytomas, pituitary neuroendocrine tumors, and primary hyperparathyroidism.
* Familial isolated NENs, including familial isolated pituitary adenoma, familial pheochromocytomas and paragangliomas, familial primary hyperparathyroidism, familial gastrointestinal stromal tumors and X-linked acrogigantism.
* Clinical syndromes encompassing NENs, with familial or sporadic presentation, including Carney complex, Carney-Stratakis syndrome, Carney triad, Cowden syndrome, DICER1 syndrome, Li-Fraumeni syndrome, Lynch syndrome, multiple endocrine neoplasia type 1, multiple endocrine neoplasia type 2, multiple endocrine neoplasia type 4, neurofibromatosis type 1, Pacak-Zhuang syndrome, paraganglioma, pheochromocytoma and pituitary adenoma syndrome, tuberous sclerosis complex, Von Hippel Lindau syndrome.

Exclusion criteria:

* Age <18 years.
* Refusal to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with new or previous clinical diagnosis of the conditions included in the eligibility criteria under follow up at either of two reference hospitals in Mexico City: Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, and Specialties Hospital of Centro Médico Nacional Siglo XXI, Instituto Mexicano del Seguro Social. All individuals must provide written informed consent to be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 750 (Estimated)
Dates: Start 2022-08-03 (Actual); Primary Completion 2037-03-01 (Estimated); Study Completion 2037-03-01 (Estimated)

PRIMARY OUTCOMES:
Detection of a germline or somatic genetic defect of interest. | Up to fifteen years from the date of recruitment.
  Detection of a genetic defect classified as pathogenic, likely pathogenic, or of uncertain significance in accordance with the criteria of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology.

CONTACTS AND LOCATIONS:
Overall Officials: Laura C Hernández Ramírez, MD, PhD, Principal Investigator — Universidad Nacional Autonoma de Mexico
Locations (3):
- Mexico (3):
  - Hospital de Especialidades, Centro Médico Nacional Siglo XXI, Instituto Mexicano del Seguro Social, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico City
  - Red de Apoyo a la Investigación, Coordinación de la Investigación Científica, Universidad Nacional Autónoma de México, Mexico City, Mexico City

REFERENCES:
- [Background] Kloppel G, Rindi G, Anlauf M, Perren A, Komminoth P. Site-specific biology and pathology of gastroenteropancreatic neuroendocrine tumors. Virchows Arch. 2007 Aug;451 Suppl 1:S9-27. doi: 10.1007/s00428-007-0461-0. Epub 2007 Aug 8. PMID 17684761
- [Background] Asa SL, Mete O, Cusimano MD, McCutcheon IE, Perry A, Yamada S, Nishioka H, Casar-Borota O, Uccella S, La Rosa S, Grossman AB, Ezzat S; Attendees of the 15th Meeting of the International Pituitary Pathology Club, Istanbul October 2019. Pituitary neuroendocrine tumors: a model for neuroendocrine tumor classification. Mod Pathol. 2021 Sep;34(9):1634-1650. doi: 10.1038/s41379-021-00820-y. Epub 2021 May 21. PMID 34017065
- [Background] Johansson E, Andersson L, Ornros J, Carlsson T, Ingeson-Carlsson C, Liang S, Dahlberg J, Jansson S, Parrillo L, Zoppoli P, Barila GO, Altschuler DL, Padula D, Lickert H, Fagman H, Nilsson M. Revising the embryonic origin of thyroid C cells in mice and humans. Development. 2015 Oct 15;142(20):3519-28. doi: 10.1242/dev.126581. Epub 2015 Sep 22. PMID 26395490
- [Background] Kulke MH, Shah MH, Benson AB 3rd, Bergsland E, Berlin JD, Blaszkowsky LS, Emerson L, Engstrom PF, Fanta P, Giordano T, Goldner WS, Halfdanarson TR, Heslin MJ, Kandeel F, Kunz PL, Kuvshinoff BW 2nd, Lieu C, Moley JF, Munene G, Pillarisetty VG, Saltz L, Sosa JA, Strosberg JR, Vauthey JN, Wolfgang C, Yao JC, Burns J, Freedman-Cass D; National comprehensive cancer network. Neuroendocrine tumors, version 1.2015. J Natl Compr Canc Netw. 2015 Jan;13(1):78-108. doi: 10.6004/jnccn.2015.0011. PMID 25583772
- [Background] Crona J, Skogseid B. GEP- NETS UPDATE: Genetics of neuroendocrine tumors. Eur J Endocrinol. 2016 Jun;174(6):R275-90. doi: 10.1530/EJE-15-0972. PMID 27165966
- [Background] Furlan A, Dyachuk V, Kastriti ME, Calvo-Enrique L, Abdo H, Hadjab S, Chontorotzea T, Akkuratova N, Usoskin D, Kamenev D, Petersen J, Sunadome K, Memic F, Marklund U, Fried K, Topilko P, Lallemend F, Kharchenko PV, Ernfors P, Adameyko I. Multipotent peripheral glial cells generate neuroendocrine cells of the adrenal medulla. Science. 2017 Jul 7;357(6346):eaal3753. doi: 10.1126/science.aal3753. PMID 28684471
- [Background] Kastriti ME, Kameneva P, Kamenev D, Dyachuk V, Furlan A, Hampl M, Memic F, Marklund U, Lallemend F, Hadjab S, Calvo-Enrique L, Ernfors P, Fried K, Adameyko I. Schwann Cell Precursors Generate the Majority of Chromaffin Cells in Zuckerkandl Organ and Some Sympathetic Neurons in Paraganglia. Front Mol Neurosci. 2019 Jan 25;12:6. doi: 10.3389/fnmol.2019.00006. eCollection 2019. PMID 30740044
- [Background] Zandee WT, Kamp K, van Adrichem RC, Feelders RA, de Herder WW. Effect of hormone secretory syndromes on neuroendocrine tumor prognosis. Endocr Relat Cancer. 2017 Jul;24(7):R261-R274. doi: 10.1530/ERC-16-0538. Epub 2017 May 8. PMID 28483790
- [Background] Melmed S. Pituitary-Tumor Endocrinopathies. N Engl J Med. 2020 Mar 5;382(10):937-950. doi: 10.1056/NEJMra1810772. No abstract available. PMID 32130815
- [Background] Yao JC, Hassan M, Phan A, Dagohoy C, Leary C, Mares JE, Abdalla EK, Fleming JB, Vauthey JN, Rashid A, Evans DB. One hundred years after "carcinoid": epidemiology of and prognostic factors for neuroendocrine tumors in 35,825 cases in the United States. J Clin Oncol. 2008 Jun 20;26(18):3063-72. doi: 10.1200/JCO.2007.15.4377. PMID 18565894
- [Background] Capdevila J, Casanovas O, Salazar R, Castellano D, Segura A, Fuster P, Aller J, Garcia-Carbonero R, Jimenez-Fonseca P, Grande E, Castano JP. Translational research in neuroendocrine tumors: pitfalls and opportunities. Oncogene. 2017 Apr 6;36(14):1899-1907. doi: 10.1038/onc.2016.316. Epub 2016 Sep 19. PMID 27641330
- [Background] Buffet A, Burnichon N, Favier J, Gimenez-Roqueplo AP. An overview of 20 years of genetic studies in pheochromocytoma and paraganglioma. Best Pract Res Clin Endocrinol Metab. 2020 Mar;34(2):101416. doi: 10.1016/j.beem.2020.101416. Epub 2020 Mar 10. PMID 32295730
- [Background] McDonnell JE, Gild ML, Clifton-Bligh RJ, Robinson BG. Multiple endocrine neoplasia: an update. Intern Med J. 2019 Aug;49(8):954-961. doi: 10.1111/imj.14394. PMID 31387156
- [Background] Chevalier B, Dupuis H, Jannin A, Lemaitre M, Do Cao C, Cardot-Bauters C, Espiard S, Vantyghem MC. Phakomatoses and Endocrine Gland Tumors: Noteworthy and (Not so) Rare Associations. Front Endocrinol (Lausanne). 2021 May 6;12:678869. doi: 10.3389/fendo.2021.678869. eCollection 2021. PMID 34025587
- [Background] Denes J, Korbonits M. The clinical aspects of pituitary tumour genetics. Endocrine. 2021 Mar;71(3):663-674. doi: 10.1007/s12020-021-02633-0. Epub 2021 Feb 4. PMID 33543431
- [Background] Pitsava G, Settas N, Faucz FR, Stratakis CA. Carney Triad, Carney-Stratakis Syndrome, 3PAS and Other Tumors Due to SDH Deficiency. Front Endocrinol (Lausanne). 2021 May 3;12:680609. doi: 10.3389/fendo.2021.680609. eCollection 2021. PMID 34012423
- [Background] Halperin R, Tirosh A. Non-Interventional Management of Advanced Pancreatic Neuroendocrine Neoplasms in Patients with von Hippel-Lindau Disease. Cancers (Basel). 2023 Mar 13;15(6):1739. doi: 10.3390/cancers15061739. PMID 36980625
- [Background] WILLIAMS ED. A REVIEW OF 17 CASES OF CARCINOMA OF THE THYROID AND PHAEOCHROMOCYTOMA. J Clin Pathol. 1965 May;18(3):288-92. doi: 10.1136/jcp.18.3.288. PMID 14304238
- [Background] Chong GC, Beahrs OH, Sizemore GW, Woolner LH. Medullary carcinoma of the thyroid gland. Cancer. 1975 Mar;35(3):695-704. doi: 10.1002/1097-0142(197503)35:33.0.co;2-w. PMID 1111937
- [Background] Fountain JW, Wallace MR, Brereton AM, O'Connell P, White RL, Rich DC, Ledbetter DH, Leach RJ, Fournier RE, Menon AG, et al. Physical mapping of the von Recklinghausen neurofibromatosis region on chromosome 17. Am J Hum Genet. 1989 Jan;44(1):58-67. PMID 2491783
- [Background] Ledbetter DH, Rich DC, O'Connell P, Leppert M, Carey JC. Precise localization of NF1 to 17q11.2 by balanced translocation. Am J Hum Genet. 1989 Jan;44(1):20-4. PMID 2491776
- [Background] Latif F, Tory K, Gnarra J, Yao M, Duh FM, Orcutt ML, Stackhouse T, Kuzmin I, Modi W, Geil L, et al. Identification of the von Hippel-Lindau disease tumor suppressor gene. Science. 1993 May 28;260(5112):1317-20. doi: 10.1126/science.8493574.
- [Background] Chandrasekharappa SC, Guru SC, Manickam P, Olufemi SE, Collins FS, Emmert-Buck MR, Debelenko LV, Zhuang Z, Lubensky IA, Liotta LA, Crabtree JS, Wang Y, Roe BA, Weisemann J, Boguski MS, Agarwal SK, Kester MB, Kim YS, Heppner C, Dong Q, Spiegel AM, Burns AL, Marx SJ. Positional cloning of the gene for multiple endocrine neoplasia-type 1. Science. 1997 Apr 18;276(5311):404-7. doi: 10.1126/science.276.5311.404. PMID 9103196
- [Background] Wells SA Jr, Asa SL, Dralle H, Elisei R, Evans DB, Gagel RF, Lee N, Machens A, Moley JF, Pacini F, Raue F, Frank-Raue K, Robinson B, Rosenthal MS, Santoro M, Schlumberger M, Shah M, Waguespack SG; American Thyroid Association Guidelines Task Force on Medullary Thyroid Carcinoma. Revised American Thyroid Association guidelines for the management of medullary thyroid carcinoma. Thyroid. 2015 Jun;25(6):567-610. doi: 10.1089/thy.2014.0335. PMID 25810047
- [Background] Iacovazzo D, Hernandez-Ramirez LC, Korbonits M. Sporadic pituitary adenomas: the role of germline mutations and recommendations for genetic screening. Expert Rev Endocrinol Metab. 2017 Mar;12(2):143-153. doi: 10.1080/17446651.2017.1306439. PMID 30063429
- [Background] Papathomas TG, Suurd DPD, Pacak K, Tischler AS, Vriens MR, Lam AK, de Krijger RR. What Have We Learned from Molecular Biology of Paragangliomas and Pheochromocytomas? Endocr Pathol. 2021 Mar;32(1):134-153. doi: 10.1007/s12022-020-09658-7. Epub 2021 Jan 12. PMID 33433885
- [Background] Jha S, Simonds WF. Molecular and Clinical Spectrum of Primary Hyperparathyroidism. Endocr Rev. 2023 Sep 15;44(5):779-818. doi: 10.1210/endrev/bnad009. PMID 36961765
- [Background] Perez-Rivas LG, Simon J, Albani A, Tang S, Roeber S, Assie G, Deutschbein T, Fassnacht M, Gadelha MR, Hermus AR, Stalla GK, Tichomirowa MA, Rotermund R, Flitsch J, Buchfelder M, Nasi-Kordhishti I, Honegger J, Thorsteinsdottir J, Saeger W, Herms J, Reincke M, Theodoropoulou M. TP53 mutations in functional corticotroph tumors are linked to invasion and worse clinical outcome. Acta Neuropathol Commun. 2022 Sep 19;10(1):139. doi: 10.1186/s40478-022-01437-1. PMID 36123588
- [Background] Lin AL, Rudneva VA, Richards AL, Zhang Y, Woo HJ, Cohen M, Tisnado J, Majd N, Wardlaw SL, Page-Wilson G, Sengupta S, Chow F, Goichot B, Ozer BH, Dietrich J, Nachtigall L, Desai A, Alano T, Ogilive S, Solit DB, Bale TA, Rosenblum M, Donoghue MTA, Geer EB, Tabar V. Genome-wide loss of heterozygosity predicts aggressive, treatment-refractory behavior in pituitary neuroendocrine tumors. Acta Neuropathol. 2024 May 17;147(1):85. doi: 10.1007/s00401-024-02736-8. PMID 38758238
- [Background] Webster AP, Thirlwell C. The Molecular Biology of Midgut Neuroendocrine Neoplasms. Endocr Rev. 2024 May 7;45(3):343-350. doi: 10.1210/endrev/bnad034. PMID 38123518
- [Background] Denes J, Swords F, Rattenberry E, Stals K, Owens M, Cranston T, Xekouki P, Moran L, Kumar A, Wassif C, Fersht N, Baldeweg SE, Morris D, Lightman S, Agha A, Rees A, Grieve J, Powell M, Boguszewski CL, Dutta P, Thakker RV, Srirangalingam U, Thompson CJ, Druce M, Higham C, Davis J, Eeles R, Stevenson M, O'Sullivan B, Taniere P, Skordilis K, Gabrovska P, Barlier A, Webb SM, Aulinas A, Drake WM, Bevan JS, Preda C, Dalantaeva N, Ribeiro-Oliveira A Jr, Garcia IT, Yordanova G, Iotova V, Evanson J, Grossman AB, Trouillas J, Ellard S, Stratakis CA, Maher ER, Roncaroli F, Korbonits M. Heterogeneous genetic background of the association of pheochromocytoma/paraganglioma and pituitary adenoma: results from a large patient cohort. J Clin Endocrinol Metab. 2015 Mar;100(3):E531-41. doi: 10.1210/jc.2014-3399. Epub 2014 Dec 12. PMID 25494863
- [Background] Xekouki P, Szarek E, Bullova P, Giubellino A, Quezado M, Mastroyannis SA, Mastorakos P, Wassif CA, Raygada M, Rentia N, Dye L, Cougnoux A, Koziol D, Sierra Mde L, Lyssikatos C, Belyavskaya E, Malchoff C, Moline J, Eng C, Maher LJ 3rd, Pacak K, Lodish M, Stratakis CA. Pituitary adenoma with paraganglioma/pheochromocytoma (3PAs) and succinate dehydrogenase defects in humans and mice. J Clin Endocrinol Metab. 2015 May;100(5):E710-9. doi: 10.1210/jc.2014-4297. Epub 2015 Feb 19. PMID 25695889
- [Background] Persani L, de Filippis T, Colombo C, Gentilini D. GENETICS IN ENDOCRINOLOGY: Genetic diagnosis of endocrine diseases by NGS: novel scenarios and unpredictable results and risks. Eur J Endocrinol. 2018 Sep;179(3):R111-R123. doi: 10.1530/EJE-18-0379. Epub 2018 Jun 7. PMID 29880707
- [Background] Seabrook AJ, Harris JE, Velosa SB, Kim E, McInerney-Leo AM, Dwight T, Hockings JI, Hockings NG, Kirk J, Leo PJ, Love AJ, Luxford C, Marshall M, Mete O, Pennisi DJ, Brown MA, Gill AJ, Hockings GI, Clifton-Bligh RJ, Duncan EL. Multiple Endocrine Tumors Associated with Germline MAX Mutations: Multiple Endocrine Neoplasia Type 5? J Clin Endocrinol Metab. 2021 Mar 25;106(4):1163-1182. doi: 10.1210/clinem/dgaa957. PMID 33367756
- [Background] Seabrook A, Wijewardene A, De Sousa S, Wong T, Sheriff N, Gill AJ, Iyer R, Field M, Luxford C, Clifton-Bligh R, McCormack A, Tucker K. MEN4, the MEN1 Mimicker: A Case Series of three Phenotypically Heterogenous Patients With Unique CDKN1B Mutations. J Clin Endocrinol Metab. 2022 Jul 14;107(8):2339-2349. doi: 10.1210/clinem/dgac162. PMID 35323929
- [Background] Thakker RV, Newey PJ, Walls GV, Bilezikian J, Dralle H, Ebeling PR, Melmed S, Sakurai A, Tonelli F, Brandi ML; Endocrine Society. Clinical practice guidelines for multiple endocrine neoplasia type 1 (MEN1). J Clin Endocrinol Metab. 2012 Sep;97(9):2990-3011. doi: 10.1210/jc.2012-1230. Epub 2012 Jun 20. PMID 22723327
- [Background] Hernandez-Ramirez LC, Gabrovska P, Denes J, Stals K, Trivellin G, Tilley D, Ferrau F, Evanson J, Ellard S, Grossman AB, Roncaroli F, Gadelha MR, Korbonits M; International FIPA Consortium. Landscape of Familial Isolated and Young-Onset Pituitary Adenomas: Prospective Diagnosis in AIP Mutation Carriers. J Clin Endocrinol Metab. 2015 Sep;100(9):E1242-54. doi: 10.1210/jc.2015-1869. PMID 26186299
- [Background] Silva-Zolezzi I, Hidalgo-Miranda A, Estrada-Gil J, Fernandez-Lopez JC, Uribe-Figueroa L, Contreras A, Balam-Ortiz E, del Bosque-Plata L, Velazquez-Fernandez D, Lara C, Goya R, Hernandez-Lemus E, Davila C, Barrientos E, March S, Jimenez-Sanchez G. Analysis of genomic diversity in Mexican Mestizo populations to develop genomic medicine in Mexico. Proc Natl Acad Sci U S A. 2009 May 26;106(21):8611-6. doi: 10.1073/pnas.0903045106. Epub 2009 May 11. PMID 19433783
- [Background] Ziyatdinov A, Torres J, Alegre-Diaz J, Backman J, Mbatchou J, Turner M, Gaynor SM, Joseph T, Zou Y, Liu D, Wade R, Staples J, Panea R, Popov A, Bai X, Balasubramanian S, Habegger L, Lanche R, Lopez A, Maxwell E, Jones M, Garcia-Ortiz H, Ramirez-Reyes R, Santacruz-Benitez R, Nag A, Smith KR, Damask A, Lin N, Paulding C, Reppell M, Zollner S, Jorgenson E, Salerno W, Petrovski S, Overton J, Reid J, Thornton TA, Abecasis G, Berumen J, Orozco-Orozco L, Collins R; Regeneron Genetics Center; Mexico City Prospective Study; Baras A, Hill MR, Emberson JR, Marchini J, Kuri-Morales P, Tapia-Conyer R. Genotyping, sequencing and analysis of 140,000 adults from Mexico City. Nature. 2023 Oct;622(7984):784-793. doi: 10.1038/s41586-023-06595-3. Epub 2023 Oct 11. PMID 37821707
- [Background] Richards S, Aziz N, Bale S, Bick D, Das S, Gastier-Foster J, Grody WW, Hegde M, Lyon E, Spector E, Voelkerding K, Rehm HL; ACMG Laboratory Quality Assurance Committee. Standards and guidelines for the interpretation of sequence variants: a joint consensus recommendation of the American College of Medical Genetics and Genomics and the Association for Molecular Pathology. Genet Med. 2015 May;17(5):405-24. doi: 10.1038/gim.2015.30. Epub 2015 Mar 5. PMID 25741868